CLINICAL TRIAL: NCT05025618
Title: Medico-economic Assessment of Adaptative Radiotherapy to Decrease Xerostomia in Locally Advanced Oropharynx Xerostomia
Brief Title: Adaptative Radiotherapy to Decrease Xerostomia in Oropharynx Carcinoma (ARTOME)
Acronym: ARTOME
Status: Completed | Type: Observational
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-7-10-002
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Oropharynx Cancer
Keywords: adaptative radiotherapy; xerostomia; medico-economic assessment
MeSH Terms: conditions — Oropharyngeal Neoplasms; Xerostomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Standard treatment for oropharynx cancer is radiotherapy by intensity modulation with only one planification before treatment. Adaptative radiotherapy integrates one or several planifications during treatment radiotherapy in order to take into account anatomic modifications that occurs.

Adaptative radiotherapy is very expensive, complex and is consuming human resources as well as equipment.

ARTIX study (NCT01874587) entitled "Phase III trial testing the benefit of intensity-modulated radiotherapy with weekly replanifications versus intensity modulated radiotherapy with only one planification in locally advanced oropharynx carcinoma for decreasing xerostomia" is completed and clinical data from this study are used to analyse if xerostomia is decreased when adaptative radiotherapy is used.

ARTOME study will assess cost-efficiency and cost utility between standard treatment (one pretherapeutic planification) and experimental treatment (weekly replanifications during treatment). Clinical data from ARTIX study will be used for ARTOME study.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced non-metastatic carcinoma of the oropharynx limited to T3 and T4 (whatever the N) and N2-N3 (whatever the T)(AJCC stage III-IV)
* Age ≥ 18 years and ≤ 75 years
* Performance status (WHO ≤ 2)
* Renal, hepatic and cardiovascular functions allowing systemic treatment administration
* Adapted stomatologic care
* Signed informed consent form
* Membership or beneficiary of a national insurance scheme

Exclusion Criteria:

* Both parotids totally included in the target volume
* Stages T1 or T2 with positive node disease N1
* Neoadjuvant chemotherapy
* Exereses of primitive tumor and/or nodes
* History of other cancer within 5 years (except for basocellular epithelioma and cervical)
* Previous neck radiotherapy
* Platinum salts, 5FluoroUracile (5FU) agents or cetuximab chemotherapy
* Unstable diseases (cardiovascular, renal, pulmonary, systemic lupus or sclerodermia) incompatible with study participation
* Patient participating in other therapeutic trial with experimental drug, 30 days before the inclusion.
* Patient already recruited in another biomedical research ( non interventional study is authorized)
* Pregnant or breast feeding patients
* Patient deprived of liberty, under tutorship, guardianship or placed under judicial protection
* Patient is deemed incapable of giving informed consent
* Patients who, for family, social, geographic or psychological reasons, cannot be adequately followed up and/or are incapable of undergoing regular controls.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for oropharynx cancer in specialized hospitals
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2013-07-05 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Cost utility analysis of standard radiotherapy (one pretherapeutic planification) compared to adaptative (weekly planification) | 2 years after end of radiotherapy treatment
  The cost utility analysis is expressed in cost per one year life gained

CONTACTS AND LOCATIONS:
Overall Officials: Renaud De Crevoisier, Professor, Principal Investigator — Centre Eugène Marquis
Locations (11):
- France (11):
  - Clinique Claude Bernard, Albi
  - Clinique Pasteur Lanroze, Brest
  - CRLCC Baclesse, Caen
  - CRLCC Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - CRLCC Antoine Lacassagne, Nice
  - CHU de la Milétrie, Poitiers
  - Centre Eugene Marquis, Rennes
  - CRLCC Henri Becquerel, Rouen
  - Centre Paul Strauss, Strasbourg
  - CHU Tours - Hôpital Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: No